CLINICAL TRIAL: NCT06491394
Title: Effect of Lactoferrin Administration on Rhabdomyolysis-induced Heart and Kidney Injury in Rats
Brief Title: Lactoferrin Effect on Kidney and Heart of Rhabdomyolysis Rats
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Asmaa Abdel-mageed Muhammed, Lecturer, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Lactoferrin in rhabdomyolysis
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Rhabdomyolysis
MeSH Terms: conditions — Rhabdomyolysis | interventions — Lactoferrin; Glycerol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control (Sham Comparator): Normal saline will be administered once to rats intramuscularly (10 mL/kg).
  Interventions: Diagnostic Test: iron; Diagnostic Test: MDA, TAC, and GSH; Diagnostic Test: Nrf2; Diagnostic Test: AMPK; Diagnostic Test: HO-1
- RM (Active Comparator): A single intramuscular injection of GLY 50% (10 mL/kg) after 24-h water deprivation and normal saline (4ml/kg) will be administered by gavage.
  Interventions: Diagnostic Test: iron; Diagnostic Test: MDA, TAC, and GSH; Diagnostic Test: Nrf2; Diagnostic Test: AMPK; Diagnostic Test: HO-1; Drug: glycerin
- Lf-RM (Active Comparator): A single intramuscular injection of GLY 50% (10 mL/kg) after 24-h water deprivation and Lf (1000 mg/kg in normal saline, volume 4 mL/kg) will be administered by gavage 30 min. before RM induction
  Interventions: Drug: Lactoferrin; Diagnostic Test: iron; Diagnostic Test: MDA, TAC, and GSH; Diagnostic Test: Nrf2; Diagnostic Test: AMPK; Diagnostic Test: HO-1; Drug: glycerin
- RM-Lf (Active Comparator): A single intramuscular injection of GLY 50% (10 mL/kg) after 24-h water deprivation and Lf (1000 mg/kg in normal saline, volume 4 mL/kg) will be administered by gavage 30 min. after RM induction.
  Interventions: Drug: Lactoferrin; Diagnostic Test: iron; Diagnostic Test: MDA, TAC, and GSH; Diagnostic Test: Nrf2; Diagnostic Test: AMPK; Diagnostic Test: HO-1; Drug: glycerin

INTERVENTIONS:
Drug: Lactoferrin — an iron-binding protein
  Arms: Lf-RM; RM-Lf
Diagnostic Test: iron — Iron in kidney and heart tissues
Diagnostic Test: MDA, TAC, and GSH — Oxidative stress levels in kidney and heart tissues
  Other Names: Malondialdehyde, Total antioxidant, and glutathione
Diagnostic Test: Nrf2 — Nrf2 expression in kidney and heart tissues
  Other Names: Nuclear factor erythroid 2-related factor 2
Diagnostic Test: AMPK — AMPK levels in heart and kidney tissues
  Other Names: Adenosine monophosphate-activated protein kinase
Diagnostic Test: HO-1 — HO-1 levels in kidney and heart tissues
  Other Names: heme oxygenase-1
Drug: glycerin — GLY intramuscular injection for rhabdomyolysis induction
  Other Names: GLY
  Arms: Lf-RM; RM; RM-Lf

SUMMARY:
This study focuses on detecting the possible beneficial effect of Lactoferrin (Lf) administration on the kidney and the heart of glycerol-induced rhabdomyolysis (RM) in rats and its relation to ferroptosis and AMPK/Nrf2/ HO-1 signalling pathway. The main questions it aims to answer are:

1. Is Lf administration 30 min. before or after RM induction in rats beneficial to kidneys and heart?
2. When administered to glycerol-induced rats, does Lf act by upregulating the AMPK/Nrf2/ HO-1 signalling pathway and inhibiting ferroptosis?

ELIGIBILITY:
Inclusion Criteria:

* • Twenty-four healthy male Wistar Albino rats weighing from 250 to 300 g

Exclusion Criteria:

* No exclusion criteria as this study is used to detect effects of drugs on experimental rats.

Ages: 10 Weeks to 12 Weeks | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Nrf2 expression | 2 months
  Nrf2 expression in heart and kidney tissues
AMPK levels | 2 months
  AMPK levels in kidney and heart tissue homogenate
HO-1 levels | 2 months
  HO-1 levels in kidney and heart tissue homogenate

SECONDARY OUTCOMES:
iron levels | 2 months
  Iron levels in heart and kidney tissue homogenate
MDA levels | 2 months
  MDA levels in heart and kidney tissue homogenate
TAC levels | 2 months
  TAC levels in heart and kidney tissue homogenate
GSH levels | 2 months
  GSH levels in heart and kidney tissue homogenate

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Aswān, Aswan Governorate, Egypt

REFERENCES:
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/32601262/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27161318/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34860639/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34091586/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35595070/